CLINICAL TRIAL: NCT06870656
Title: Muscle Isometric Contraction for the Treatment of Knee Osteoarthritis
Acronym: KOA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Sport University (Other)
Responsible Party: Principal Investigator, Cheng Liang, Director, Chengdu Sport University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Muscle isometric contraction; 2024ZYD0001 (Other Grant/Funding Number: This work was supported by the Central Guidance for Local Science and Technology Development Fund Projects)
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis (Knee OA)
Keywords: KOA; Muscle isometric contraction
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Isometric Contraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low-intensity group (Experimental): Firstly, they received the same health education as the control group. Subsequently, the elderly individuals with Knee Osteoarthritis (KOA) underwent five interventions per week targeting the quadriceps femoris muscle. For each intervention, the quadriceps performed an isometric contraction and relaxation for 1 second each. The intervention consisted of 10 repetitions per set of Muscle Isometric Contraction (MIC), guided by a rhythmic timer, for a total of 10 sets, with a 30-second rest between sets. The entire intervention lasted for 16 weeks.
  Interventions: Other: Low-intensity group
- Medium-intensity group (Experimental): Firstly, they received the same health education as the control group. Subsequently, the elderly individuals with Knee Osteoarthritis (KOA) underwent five interventions per week targeting the quadriceps femoris muscle. For each intervention, the quadriceps performed an isometric contraction and relaxation for 1 second each. The intervention consisted of 20 repetitions per set of Muscle Isometric Contraction (MIC), guided by a rhythmic timer, for a total of 10 sets, with a 30-second rest between sets. The entire intervention lasted for 16 weeks.
  Interventions: Other: Medium-intensity group
- High-intensity group (Experimental): Firstly, they received the same health education as the control group. Subsequently, the elderly individuals with Knee Osteoarthritis (KOA) underwent five interventions per week targeting the quadriceps femoris muscle. For each intervention, the quadriceps performed an isometric contraction and relaxation for 1 second each. The intervention consisted of 30 repetitions per set of Muscle Isometric Contraction (MIC), guided by a rhythmic timer, for a total of 10 sets, with a 30-second rest between sets. The entire intervention lasted for 16 weeks.
  Interventions: Other: High-intensity group
- Control group (No Intervention): Health Education: All participants received standardized health guidance, which was delivered in the form of a weekly 60-minute lecture. The content of the lectures included the following:
  Emphasizing the importance of close cooperation with medical professionals for maintaining health.
  Explaining the etiology, progression, and treatment options for Knee Osteoarthritis (KOA).
  Discussing the positive impact of family and social support on recovery. Providing guidance on establishing healthy daily living habits, such as protecting the affected knee joints, avoiding prolonged walking, climbing, or frequent use of stairs, and correcting poor postures (e.g., prolonged standing, kneeling, and squatting).
  For those who are overweight, weight loss was recommended.

INTERVENTIONS:
Other: Low-intensity group — Firstly, they received the same health education as the control group. Subsequently, the elderly individuals with Knee Osteoarthritis (KOA) underwent five interventions per week targeting the quadriceps femoris muscle. For each intervention, the quadriceps performed an isometric contraction and relaxation for 1 second each. The intervention consisted of 10 repetitions per set of Muscle Isometric Contraction (MIC), guided by a rhythmic timer, for a total of 10 sets, with a 30-second rest between sets. The entire intervention lasted for 16 weeks.
  Other Names: Muscle Isometric Contraction
  Arms: Low-intensity group
Other: Medium-intensity group — Firstly, they received the same health education as the control group. Subsequently, the elderly individuals with Knee Osteoarthritis (KOA) underwent five interventions per week targeting the quadriceps femoris muscle. For each intervention, the quadriceps performed an isometric contraction and relaxation for 1 second each. The intervention consisted of 20 repetitions per set of Muscle Isometric Contraction (MIC), guided by a rhythmic timer, for a total of 10 sets, with a 30-second rest between sets. The entire intervention lasted for 16 weeks.
  Arms: Medium-intensity group
Other: High-intensity group — Firstly, they received the same health education as the control group. Subsequently, the elderly individuals with Knee Osteoarthritis (KOA) underwent five interventions per week targeting the quadriceps femoris muscle. For each intervention, the quadriceps performed an isometric contraction and relaxation for 1 second each. The intervention consisted of 30 repetitions per set of Muscle Isometric Contraction (MIC), guided by a rhythmic timer, for a total of 10 sets, with a 30-second rest between sets. The entire intervention lasted for 16 weeks.
  Arms: High-intensity group

SUMMARY:
This study compares the effects of three different intensities of Muscle Isometric Contraction (MIC) on balance ability, proprioception, muscle strength, KOA symptoms, and inflammatory factors in synovial fluid among elderly individuals with Knee Osteoarthritis (KOA).

DETAILED DESCRIPTION:
A total of 120 elderly individuals with Knee Osteoarthritis (KOA) will be recruited and randomly assigned into four groups using a digital randomization method: low-intensity group (n = 30), medium-intensity group (n = 30), high-intensity group (n = 30), and control group (n = 30). The elderly individuals in the low-, medium-, and high-intensity groups will receive five interventions per week targeting the quadriceps femoris muscle. For each intervention, the quadriceps will perform an isometric contraction and relaxation for 1 second each. The low-, medium-, and high-intensity groups will perform 10, 20, and 30 repetitions per set, respectively, of Muscle Isometric Contraction (MIC) (guided by a rhythmic timer), completing a total of 10 sets with a 30-second rest between sets. The entire intervention will last for 16 weeks. Researchers will follow up with participants weekly to complete exercise record forms, ensuring that all subjects maintain their original lifestyle and dietary habits. The study aims to compare the effects of three different intensities of MIC on balance ability, proprioception, muscle strength, KOA symptoms, and inflammatory factors in synovial fluid among elderly individuals with KOA.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 60 to 80 years;
* Based on the diagnostic criteria for knee osteoarthritis (KOA) established by the American College of Rheumatology in 2001, participants with KOA graded 1 to 3 were selected;
* Compliance with the Declaration of Helsinki and signing of the informed consent form.

Exclusion Criteria:

* Cardiovascular diseases;
* Need for surgery or pharmacological treatment in the near future;
* Neuromuscular diseases;
* Currently engaged in regular exercise.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
KOA Symptoms | 16 weeks
  The symptoms of patients with Knee Osteoarthritis (KOA) were assessed using the Western Ontario and McMaster Universities Arthritis Index (WOMAC) scale. This scale comprises three dimensions: pain (5 items), stiffness (2 items), and functional limitation (17 items), totaling 24 items. Participants were required to mark their responses on a visual analog scale ranging from 0 to 100 millimeters, which were then measured and recorded by professionals using a ruler. The maximum scores for pain, stiffness, and functional limitation are 500, 200, and 1700 points, respectively. Higher scores indicate greater severity of symptoms. For the Chinese KOA patient population, the scale has demonstrated high internal consistency (Cronbach's α > 0.7) and good reliability (ICC > 0.8) (Xie et al., Quality of Life Research, 2008).
Balance Ability | 16 weeks
  The BioDex Balance System from the United States was used to test the participants' balance ability, with three tests conducted and the average value taken.
Muscle Strength | 16 weeks
  The IsoMed 2000 isokinetic dynamometer from Germany was used to test the isokinetic muscle strength of the participants' bilateral knee joints.
Proprioception | 16 weeks
  The BioDex isokinetic dynamometer from the United States was used to test the proprioception of the participants' dominant knee joint.
Expression of IL-1β in Knee Synovial Fluid | 16 weeks
  Synovial fluid was aspirated from one or both knee joints of the participants, with a total volume of 1 mL collected. The expression of IL-1β mRNA was measured using RT-qPCR.
Expression of TNF-α in Knee Synovial Fluid | 16 weeks
  Synovial fluid was aspirated from one or both knee joints of the participants, with a total volume of 1 mL collected. The expression of TNF-α mRNA was measured using RT-qPCR.
Expression of MMP-13 in Knee Synovial Fluid | 16 weeks
  Synovial fluid was aspirated from one or both knee joints of the participants, with a total volume of 1 mL collected. The expression of MMP-13 mRNA was measured using RT-qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Cheng, Principal Investigator — Chengdu Sport University

IPD SHARING:
Plan to Share IPD: No